CLINICAL TRIAL: NCT04194957
Title: Improving the Safety of Fluoropyrimidine-based Chemotherapy by Combined DPYD Genotype-guided and DPD Phenotype-guided Dose Individualization: The ALPE2U Study
Brief Title: Improving the Safety of Fluoropyrimidine-based Chemotherapy
Acronym: Alpe2U
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M19ALP
Record Dates: First submitted 2019-11-15; First posted 2019-12-11 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Neoplasms
Keywords: Fluoropyrimidines; Phenotyping; Genotyping; Dose-individualization; Capecitabine; 5-Fluorouracil; 5-FU
MeSH Terms: conditions — Neoplasms | interventions — Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Wild type for DPYD (Experimental): Patients screened for four single nucleotide polymorphisms (SNPs) in DPYD (DPYD*2A, c.2846A>T, c.1236G>A/HapB3 and DPYD*13) that are found to be wild type for these SNPs
  Interventions: Drug: Fluoropyrimidine (capecitabine or 5-fluorouracil)
- heterozygous carrier of c.1236G>A or c.2846A>T DPYD variant (Experimental): Patients screened for four single nucleotide polymorphisms (SNPs) in DPYD (DPYD*2A, c.2846A>T, c.1236G>A/HapB3 and DPYD*13) that are found to be heterozygous for c.1236G>A or c.2846A>T of these SNPs
  Interventions: Drug: Fluoropyrimidine (capecitabine or 5-fluorouracil)
- Homozygous or compound heterozygous carrier of DPYD variants (Experimental): Patients screened for four single nucleotide polymorphisms (SNPs) in DPYD (DPYD*2A, c.2846A>T, c.1236G>A/HapB3 and DPYD*13) that are found to be homozygous or compound heterozygous for these SNPs
  Interventions: Drug: Fluoropyrimidine (capecitabine or 5-fluorouracil)

INTERVENTIONS:
Drug: Fluoropyrimidine (capecitabine or 5-fluorouracil) — Patients that are found to be wild type and have a pre-treatment uracil concentration above 16 ng/mL will receive a reduced dosage of capecitabine or 5-fluorouracil (50% reduction). The dose will be titrated after 2 cycles , to achieve maximal safe exposure. Patients that are wildtype with a uracil concentration below 16 ng/mL will receive a normal (full) dose.
  Arms: Wild type for DPYD
Drug: Fluoropyrimidine (capecitabine or 5-fluorouracil) — Patients that are heterozygous carriers of c.1236G>A or c.2846A>T DPYD variant will receive a reduced dosage of capecitabine or 5-FU (50 % reduction). The dose will be titrated after 2 cycles, to achieve maximal safe exposure.
  Arms: heterozygous carrier of c.1236G>A or c.2846A>T DPYD variant
Drug: Fluoropyrimidine (capecitabine or 5-fluorouracil) — Patients with homozygous or compound heterozygous DPYD variants will be treated with a reduced dose of capecitabine or 5-FU based on the DPD enzyme activity measured in peripheral blood mononuclear cells.
  Arms: Homozygous or compound heterozygous carrier of DPYD variants

SUMMARY:
In this study it will be determined whether the rate of severe toxicity associated with fluoropyrimidine treatment (capecitabine or 5-fluorouracil) can be significantly diminished by individualized dosing of fluoropyrimidines based on upfront phenotypic assessment of dihydropyrimidine dehydrogenase (DPD) deficiency.

DETAILED DESCRIPTION:
In this study a phenotypic approach will be studied to determine the additional value of pretreatment uracil level-guided dose individualization in wildtype patients. Patients with a pretreatment serum uracil concentration above 16 ng/ml will be treated with a 50% reduced fluoropyrimidine starting dose. The pretreatment serum uracil levels in DPYD variant carriers will be assessed retrospectively and non-interventional. Additionally, the effect of a higher dose reduction in c.1236G>A and c.2846A>T DPYD variants carriers (50% instead of 25%) will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed malignancy for which treatment with a fluoropyrimidine is considered to be in the patient's best interest
2. Patient need to be of Western descent
3. Age ≥ 18
4. Able and willing to give written informed consent
5. WHO performance status of 0, 1 or 2
6. Able and willing to undergo extra blood sampling for study related analysis
7. Adequate baseline patient characteristics, in the opinion of the treating physician (complete blood count, hepatic function which involves serum bilirubin, AST, ALT, and renal function)

Exclusion Criteria:

1. Prior treatment with fluoropyrimidines
2. Patients with known substance abuse, psychotic disorders, and/or other diseases expected to interfere with study or the patient's safety in the opinion of the treating physician
3. Patients treated with the combination of a fluoropyrimidine and irinotecan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Safety: incidence of severe fluoropyrimidine-related toxicity (CTCAE grade 3 to 5) in wild type patients | Patients with a pre-treatment uracil concentration above 16 ng/ml will be followed until end of treatment (expected average of 1 year). Otherwise, patients will be followed for the first 2 cycles (each cycle is 28 days).

SECONDARY OUTCOMES:
Safety: incidence of severe treatment-related toxicity (CTCAE grade 3 to 5) in heterozygous carriers of c.1236G>A or c.2846A>T DPYD variants | Patients will be followed during fluoropyrimidine treatment, expected average of 1 year
Assessment of pharmacokinetics: Such profile parameters will include Cmax, Tmax, AUC and elimination half-life | During the first administration of fluoropyrimidine treatment
Cost-effectiveness: medical costs that are made during fluoropyrimidine treatment seen from a health care perspective | Patients will be followed during fluoropyrimidine treatment, expected average of 1 year
Assessment of feasibility of dose titration following an initial dose reduction | During fluoropyrimidine treatment, expected average of 1 year
Assessment of geriatric parameters for grade 3-5 toxicity and/or treatment discontinuation | During fluoropyrimidine treatment, expected average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Annemieke Cats, MD, PhD, Principal Investigator — Netherlands Cancer Institute - Antoni van Leeuwenhoek
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henricks LM, Lunenburg CATC, de Man FM, Meulendijks D, Frederix GWJ, Kienhuis E, Creemers GJ, Baars A, Dezentje VO, Imholz ALT, Jeurissen FJF, Portielje JEA, Jansen RLH, Hamberg P, Ten Tije AJ, Droogendijk HJ, Koopman M, Nieboer P, van de Poel MHW, Mandigers CMPW, Rosing H, Beijnen JH, Werkhoven EV, van Kuilenburg ABP, van Schaik RHN, Mathijssen RHJ, Swen JJ, Gelderblom H, Cats A, Guchelaar HJ, Schellens JHM. DPYD genotype-guided dose individualisation of fluoropyrimidine therapy in patients with cancer: a prospective safety analysis. Lancet Oncol. 2018 Nov;19(11):1459-1467. doi: 10.1016/S1470-2045(18)30686-7. Epub 2018 Oct 19. PMID 30348537
- [Derived] Knikman JE, Gelderblom H, Beijnen JH, Cats A, Guchelaar HJ, Henricks LM. Individualized Dosing of Fluoropyrimidine-Based Chemotherapy to Prevent Severe Fluoropyrimidine-Related Toxicity: What Are the Options? Clin Pharmacol Ther. 2021 Mar;109(3):591-604. doi: 10.1002/cpt.2069. Epub 2020 Nov 12. PMID 33020924